CLINICAL TRIAL: NCT05571306
Title: Can Diabetes Distress be Reduced by Improving Entry to Care for People With Type 2 Diabetes Mellitus: A Cluster-randomized Trial
Brief Title: Can Diabetes Distress be Reduced by Improving Entry to Care for Type 2 Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11.562
Record Dates: First submitted 2022-09-28; First posted 2022-10-07 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes; Diabetes Distress
Keywords: Diabetes Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: As the study is a cluster randomized trial, General Practitioners are those being allocated for either intervention or control (care as usual), with controls being enrolled as late intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients are blinded to what treatment their are given and the investigator and outcome Assessor is likewise blinded as each patients and general practices are annonymized..
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receives a three month intervention.
  Interventions: Other: four core components care
- Care as usual (No Intervention): This arm is given care as usual provided at a General Practice in Denmark.

INTERVENTIONS:
Other: four core components care — The intervention progresses throughout the first three months for the recently diagnosed T2DM patients and is divided into four core components: 1) Improve of cross-sectoral communication and information sharing, 2) ensure systematism in care, 3) guarantee participation at a "one-stop-shop" and a start-up conversation at the municipality, and 4) improve patients coping skills.
  Other Names: Entry to care
  Arms: Intervention

SUMMARY:
Care recommendations for type 2 diabetes mellitus (T2DM) patients are clearly defined in Danish clinical guidelines: patients are offered three consultations with the general practice (GP), patients must be referred for a municipal start-up conversation, and cross-sectoral collaboration is vital to succeeding in the treatment of T2DM patients. This framework is often reported as inadequate by the patients, which increases the risk of high levels of diabetes distress (DD). Diabetes distress is the burden of living with T2DM and is associated with deleterious physical and mental health outcomes, including poor glycemic control, recurved wellbeing, and increased all-course mortality.

This project evaluates the efficacy of an entry-to-care intervention, seeking to strengthen and structure the cross-sectoral collaboration, targeting DD in people recently diagnosed with T2DM.

Intervention The intervention progresses throughout the first three months of the diagnosis. It is divided into core components: Improvements of cross-sectoral communication and information sharing, ensure systematism in care, guarantee participation at a "one-stop-shop" and a start-up conversation at the municipal, and improve patients coping skills.

Research plan This cluster-randomized control trial is conducted in the Region of Southern Denmark, with each GP randomly assigned to intervention or control. Changes in DD are the primary outcome. Data will be collected through an electronic questionnaire at baseline and 4, 12 months after diagnosis.

Perspective and expected outcomes A decrease in DD levels causes; higher level of self-care, quality of life, self-management, glycemic control and decrease the risk of severe complications and all-cause mortality. The intervention will be extrapolated to other patient groups where cross-sectoral collaboration is part of the care, increasing the treatment for these patient groups as well.

DETAILED DESCRIPTION:
1. Background When diagnosed with type 2 diabetes mellitus (T2DM), patients face numerous challenges such as emotional reactions to the diagnosis, acquiring new knowledge to better comprehend the disease, management of the disease, altering of diet, fear of complications, and potentially disrupted relationships with family and friends. To support these patients, care recommendations are clearly defined in the clinical guidelines for the treatment of T2DM (1,2). It is suggested that three consultations with the general practice (GP) are adequate to provide the patient with information about the disease, disease management, and treatment. Moreover, patients are recommended to be referred for health-education programs, lifestyle interventions, and complication screenings (1). However, it has been reported that a large proportion of patients are in fact not referred to these programs, in the municipalities, even though they explicitly wanted to (3). Also, the continuity of care and cross-sectoral collaboration between sectors have been reported to be deficient, with patients requesting more cross-sectoral collaboration and information sharing (4). These shortcomings in the organizational structure of diabetes care may result in psychological or psychosocial complications such as depression and/or diabetes-related distress (DD) Diabetes distress is the most prevalent complication in T2DM patients, with 36% reporting high or severe levels of DD (5,6). Diabetes distress refers to the negative emotional experiences resulting from receiving the disease and the challenges of living with diabetes in day-to-day activities. DD is positively associated with glycemic control and self-care, increasing the risk of complications and the higher the level of DD (7).

   Additionally, recent studies point towards an association between high levels of DD and increased mortality rate among men (8). Thus, it is of immense importance to address DD timely to prevent/reduce further exacerbation, which might lead to more severe complications. Hence, this project evaluates a structural entry-to-care intervention, created by Steno Diabetes Centre Odense (SDCO), aiming at increasing the cross-sectoral collaboration and structuring of the treatment of the first three months when diagnosed, while reducing DD among recently diagnosed T2DM patients. The intervention will facilitate cross-sectoral collaboration, provide novel, data-driven individualized recommendations to GPs, guidelines, and checklists for patients, and inclusion of the "one-stop-shop".
2. Design and Methods A: Design The design is a cluster-randomized, controlled trial conducted in the primary- and secondary sectors in the Region of Southern Denmark. It is designed to examine the effect of a structured start-up routine on recently diagnosed T2DM patients. GP will be randomly allocated to either intervention or control.

B: Intervention The intervention progresses throughout the first three months for the recently diagnosed T2DM patients and is divided into four core components: 1) Improve of cross-sectoral communication and information sharing, 2) ensure systematism in care, 3) guarantee participation at a "one-stop-shop" and a start-up conversation at the municipality, and 4) improve patients coping skills.

B1. Improve cross-sectoral communication and information sharing To increase cross-sectoral communication and information sharing, meetings between GP, municipalities, and regional hospitals will be facilitated by SDCO. Based on previous reports by SDCO, patients did not experience satisfactory cross-sectoral collaboration as part of their treatment; indeed, coherence of treatment was for some patients non-existing. Coherence to treatment has a positive and negative association with DD severity (6). Hence, the cross-sectoral meetings include knowledge sharing concerning the specific healthcare services each sector provides regarding the treatment/care of the recently diagnosed T2DM patients.

These elements are expected to increase the cross-sectoral collaboration, thus increasing care coherence felt by the patients.

B2. Systematism in care To ensure systematism and uniformity in the care given to all recently diagnosed T2DM patients, clear guidelines (developed from present recommendations by SDCO) are given to each GP (Appendix 3 Guidelines for general practice). The guidelines act as a framework of what advisable information patients are to be given at the first four consultations. Additionally, each GP is invited to an individual meeting with SDCO, where requirements and needs are discussed, thus tailoring the implementation to each GPs individual needs.

B3. A "one-stop-shop" and a start-up conversation at the municipality The report mentioned in B1 further stated that GP failed to refer patients for the start-up conversation at the municipalities, either because the GP was unaware of the proposal or due to them being uncertain of the 'service' quality. It is known that levels of DD improve if patients participate in health-related education (6), thus it is of great importance that GP does refer patients for a start-up conversation in the municipality, as they are delivering these education programs. Hence, GP must refer all patients for a start-up conversation at the municipality and for a "one-stop-shop" (an opportunity for patients to complete several required examinations e.g., blood samples, blood pressure measurement, eye, and feet screening during one appointment). These referrals do ensure automatization in the treatment of T2DM, and it provides the patients with the premises of improved care.

B4. Improvements of patients coping skills Patient information material has been developed by SDCO in collaboration with TD2M patients. This provides the patients with a greater sense of coherence, structure, and overview of the first period with their new disease and consists of 1) a checklist, ensuring that patients are given the mandatory information concerning any question they might have (Appendix 4 Checklist for patients), 2) a graphical guide throughout the first period with the disease (Flowchart of patient flow - the same as above), and 3) basic information about the disease (Steno Pjece Quick guide - Danish version). All material is designed to support the patients in the uncertainty right after the diagnosis and thus, providing them a greater understanding and transparency of the disease which in turn should minimize the levels of DD by increasing their coping skills.

C Method This project evaluates the effects of a structural entry-to-care intervention compared to usual in its ability to reduce DD among recently diagnosed T2D patients (Appendix 5 Flow of randomization) SDCO is responsible for the recruitment of GPs within the Region of Southern Denmark. GPs agreeing upon participation will be randomized for intervention or control clusters with a 1:1 allocation ratio using a random computer-generated block size of six (9).

GPs are stratified into two groups, the first including GPs with one or two capacities and the second with three or more capacities. GPs included in the 'digital individualized and collaborative treatment of T2DM in general practice' (DICTA) intervention will be excluded, thus minimizing contamination between interventions. This study requires 32 clusters (16/arm) to achieve 80% power and a 5% significance cut-off, with 270 patients required. GP recruitment occurred from May-Dec 2022. Patient recruitment is ongoing from May 2022 to Aug 2023. GPs were randomized 1:1 using computer-generated blocks of six.. Patients included must be 18+ years, understand Danish, and be diagnosed according to Danish guidelines. The intervention group will receive a three-month individualized treatment, while the control receives treatment as usual.

D Effect Evaluation The outcomes displayed below were chosen as they are validated tools measuring their area of capability and have all been validated in Danish.

D1. Primary outcome (measured at baseline, 4, and 12 months) (appendix 6 measure overview).

• Changes in DD levels measured using the diabetes distress scale (DDS) (10). The DDS scale was designed to measure the level of diabetes-related distress and potential contributing factors such as 'physician-related distress', 'regimen-related distress' etc.. Diabetes distress was chosen as the primary outcome due to it being associated with several health indicators such as the level of self-care (diet, exercise, etc.), quality of life, self-management, HbA1c, blood lipids, depression, severe complications, and all-cause mortality.

D2. Secondary outcomes (measured at baseline, 4, and 12 months)

* Improvements in the perceived quality of care will be measured through self-made questions
* Improvements in self-management measured by the Patient Activation Measure as positively related to health outcomes such as HbA1c, lipids, and blood pressure (11)
* Improvements in quality of life will be measured using the 12-item short-form survey (12). This was chosen as a measure that is comparable with the Danish population
* Improvements in self-care measured using the Summary of Diabetes Self-Care Activities Measurement (13) was chosen as self-care has been reported to be positively associated with DD
* Improvements in the clinical components HbA1c, blood pressure, blood lipids, and EKG is to be measured.

D3. Tertiary outcome Levels of depression and stress measured by the Major Depression Inventory (14) and the 2-item Stress Scale (15), respectively as patients with a higher level of depression and stress have increased levels of DD (16), therefore a planned examination of the association between depression, stress, and DD at baseline, 4, and 12 months follow-up will be conducted. Additionally, the level of social support measured using the Lubben Social Network Scale and the level of resilience measured using the Conner-Davidson Resilience Scale will likewise be compared with the levels of DD at the same time point as higher perceived social support and resilience have been reported to be associated with lower DD levels.

D4. Potential covariates including sex, age, nationality, clinical and biochemical measures, education status, marital status, comorbidity, smoking, physical activity, employment status, depression, social network, and sleep quantity and quality.

Patient-reported outcomes will be collected through an electronic survey distributed individually to the patients' e-Boks (19). Clinical and biochemical measures, such as blood pressure and HbA1c, will be collected through the clinical laboratory information system (20), and clinical biochemistry departments. These data will be linked to sociodemographic data via Statistics Denmark.

E Sample size The total number of clusters needed is calculated based on means and standard deviations from previous studies (21). A low cluster interclass correlation (0.1) and a mean group cluster size of 8 (the total number of T2DM patients each capacitate observe per year) in both the control and intervention group is expected. With a power of 80%, a dropout rate of 20%, and a significance level of 5%, 64 clusters (32 In each) and 512 patients are required for the analysis.

F Data analysis All analyses will be performed as intention-to-treat (22). The Generalized Estimating Equations model (GEE) will be used for the analysis, taking the cluster randomization into account. The model will be adjusted for the main potential confounders. The GEE analysis will be performed using STATA/BE (Version 17). The level of statistical significance will be P < 0.05. To support future hypotheses, several ad-hoc analyses will be conducted as required.

G Limitations The requirement that patients must understand Danish excludes individuals which previously have been reported to have the highest level of DD (6) and who potentially would benefit most from the intervention.

This project mainly consists of patient-reported outcomes, which increases the risk of drop-out due to the length of the questionnaire.

Clinical outcomes might not provide notable changes before two years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Understand Danish
* Diagnosed according to Danish guidelines

Exclusion Criteria:

* General Practitioners enrolled for the DD2 project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Diabetes Distress levels | measured at baseline, 4, and 12 months
  Changes in DD levels measured using the diabetes distress scale (DDS). The DDS scale was designed to measure the level of diabetes-related distress and potential contributing factors such as 'physician-related distress', 'regimen-related distress' etc..

SECONDARY OUTCOMES:
Quality of Care reported by the patients | measured at baseline, 4, and 12 months
  Changes in the perceived quality of care will be measured through self-made questions.
Changes in Self-management measured by the Patient Activation Measure questionnaire | measured at baseline, 4, and 12 months
  Changes in self-management measured by the Patient Activation Measure
Changes in the SF-12 (Quality of life) | measured at baseline, 4, and 12 months
  Changes quality of life will be measured using the 12-item short-form survey. This was chosen as a measure that is comparable with the Danish population
Changes in Self-care measured using the Summary of Diabetes Self-Care Activities Measurement questionnaire | measured at baseline, 4, and 12 months
  Changes in self-care measured using the Summary of Diabetes Self-Care Activities Measurement was chosen as self-care has been reported to be positively associated with DD
Changes in HbA1c | measured at baseline, 4, and 12 months
  Changes in HbA1c will be measured in mmol/l
Changes in Blood pressure | Measured at baseline, 4, and 12 months
  Changes in systolic and diastolic blood pressure will be measured in mmHg.
Changes in Blood lipds | Measured at baseline, 4, and 12 months
  Changes in low-density lipoprotein (LDL) and high-density lipoprotein (HDL) will be measured.

OTHER OUTCOMES:
Changes in Stress scale | measured at baseline, 4, and 12 months
  Level of stress measured by the 2-item Stress Scale
Changes in Major Depression Inventory | measured at baseline, 4, and 12 months
  Level of depression measured by the Major Depression Inventory
Changes in Social Network scale | measured at baseline, 4, and 12 months
  The level of social support measured using the Lubben Social Network Scale
Changes in Resilience measured using the Conner-Davidson Resilience Scale | measured at baseline, 4, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens Søndergaard, Phd, Principal Investigator — Research Unit of General Practice (University of Southern Denmark)
Locations (1):
- University of Soutern Denmark, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to legal issues this will for now not be available.

REFERENCES:
- [Background] Perrin NE, Davies MJ, Robertson N, Snoek FJ, Khunti K. The prevalence of diabetes-specific emotional distress in people with Type 2 diabetes: a systematic review and meta-analysis. Diabet Med. 2017 Nov;34(11):1508-1520. doi: 10.1111/dme.13448. Epub 2017 Aug 31. PMID 28799294
- [Background] Skinner TC, Joensen L, Parkin T. Twenty-five years of diabetes distress research. Diabet Med. 2020 Mar;37(3):393-400. doi: 10.1111/dme.14157. Epub 2019 Oct 31. PMID 31638279
- [Background] Peimani M, Nasli-Esfahani E, Sadeghi R. Patients' perceptions of patient-provider communication and diabetes care: A systematic review of quantitative and qualitative studies. Chronic Illn. 2020 Mar;16(1):3-22. doi: 10.1177/1742395318782378. Epub 2018 Jun 12. No abstract available. PMID 29895167
- [Background] Hayashino Y, Okamura S, Tsujii S, Ishii H; Diabetes Distress and Care Registry at Tenri Study Group. Association between diabetes distress and all-cause mortality in Japanese individuals with type 2 diabetes: a prospective cohort study (Diabetes Distress and Care Registry in Tenri [DDCRT 18]). Diabetologia. 2018 Sep;61(9):1978-1984. doi: 10.1007/s00125-018-4657-4. Epub 2018 Jun 8. PMID 29947921
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Schmitt A, Reimer A, Kulzer B, Haak T, Ehrmann D, Hermanns N. How to assess diabetes distress: comparison of the Problem Areas in Diabetes Scale (PAID) and the Diabetes Distress Scale (DDS). Diabet Med. 2016 Jun;33(6):835-43. doi: 10.1111/dme.12887. Epub 2015 Sep 8. PMID 26287511
- [Background] Sacks RM, Greene J, Hibbard J, Overton V, Parrotta CD. Does patient activation predict the course of type 2 diabetes? A longitudinal study. Patient Educ Couns. 2017 Jul;100(7):1268-1275. doi: 10.1016/j.pec.2017.01.014. Epub 2017 Jan 25. PMID 28159442
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Littman AJ, White E, Satia JA, Bowen DJ, Kristal AR. Reliability and validity of 2 single-item measures of psychosocial stress. Epidemiology. 2006 Jul;17(4):398-403. doi: 10.1097/01.ede.0000219721.89552.51. PMID 16641618
- [Background] Yang QQ, Sun JW, Shao D, Zhang HH, Bai CF, Cao FL. The Association between Diabetes Complications, Diabetes Distress, and Depressive Symptoms in Patients with Type 2 Diabetes Mellitus. Clin Nurs Res. 2021 Mar;30(3):293-301. doi: 10.1177/1054773820951933. Epub 2020 Aug 17. PMID 32799656
- [Background] Glasgow RE, Kurz D, King D, Dickman JM, Faber AJ, Halterman E, Woolley T, Toobert DJ, Strycker LA, Estabrooks PA, Osuna D, Ritzwoller D. Twelve-month outcomes of an Internet-based diabetes self-management support program. Patient Educ Couns. 2012 Apr;87(1):81-92. doi: 10.1016/j.pec.2011.07.024. Epub 2011 Sep 15. PMID 21924576
- [Background] McCoy CE. Understanding the Intention-to-treat Principle in Randomized Controlled Trials. West J Emerg Med. 2017 Oct;18(6):1075-1078. doi: 10.5811/westjem.2017.8.35985. Epub 2017 Sep 18. PMID 29085540
- [Derived] Hansen SH, Jensen TM, Petersen GS, Pouwer F, Larrabee Sonderlund A, Sondergaard J. Effect of an entry-to-care intervention on diabetes distress in individuals with newly diagnosed type 2 diabetes: a study protocol for a cluster-randomized trial. Trials. 2024 Mar 21;25(1):207. doi: 10.1186/s13063-024-07949-6. PMID 38515146
- See also: The cross-sectoral course programme for patients with type 2 diabetes - Region of Southern Jutland. — https://faelleskommunalsundhed.dk/wp-content/uploads/edagsorden-documents/5957df2f-4f19-4b95-91bf-8cad019e8892.pdf
- See also: The Danish diabetes association with a report on the life with type 2 diabetes — https://diabetes.dk/media/ql2mc4q0/rapport_livet-med-diabetes_2019.pdf
- See also: The national research centre on welfare with a report on the life with type 2 diabetes — https://www.vive.dk/da/udgivelser/livet-med-type-2-diabetes-16337/
- See also: National Knowledge Centre on Dementia and information about the outcome Major Depression Inventory — https://videnscenterfordemens.dk/da/major-depression-inventory-mdi
- See also: Description of the LSNS outcome measure. — http://www.bc.edu/bc-web/schools/ssw/sites/lubben/description.html
- See also: Description of the CD-RISC outcome measure. — https://www.cd-risc.com/
- See also: Information about e-Boks — http://www.e-boks.com/danmark/da/hvad-er-e-boks/
- See also: Where the clinical results are recieved. — http://www.cgi.com/dk/da/solutions/laboratorielosning